CLINICAL TRIAL: NCT02133638
Title: Sevoflurane-based Volatile Induction and Maintenance of Anaesthesia (VIMA) Strategy Decreases the Risk of Postoperative Delirium in Elderly Patients With Registered Cerebral Hypoxemia Episodes During General Surgery
Brief Title: Sevoflurane Decreases the Risk of Postoperative Delirium After Cerebral Hypoxemia During Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Negovsky Reanimatology Research Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sev003; s100b (Other: s100b)
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Cerebral Hypoxia; Postoperative Delirium
Keywords: Delirium; Hypoxic Brain Damage; Propofol; S100b protein; Sevoflurane
MeSH Terms: conditions — Hypoxia, Brain; Emergence Delirium; Delirium | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Active Comparator): Sevoflurane Based Volatile Induction and Maintenance of Anaesthesia
  Interventions: Drug: Sevoflurane
- Propofol (Active Comparator): Propofol Based Total Intravenous Anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Induction of anesthesia: fentanyl 2 µg kg-1 and a bolus inhalation of 8% sevoflurane in an 8 L.min-1 fresh gas flow. Anesthesia maintenance: 1 minimal alveolar concentration (MAC) sevoflurane at a low fresh gas flow of 0.6-0.8 L min-1 in a 60% air-oxygen mixture supplemented with boluses of fentanyl.
  Other Names: Sevorane; Ultane; Fluoromethyl hexafluoroisopropyl ether
  Arms: Sevoflurane
Drug: Propofol — Induction of anesthesia: propofol 2 mg kg-1 and fentanyl 4 µg kg-1. Maintenance of anesthesia: infusion of propofol 8 mg kg-1 h-1 and boluses of fentanyl 3 µg kg-1.
  Other Names: Diprivan; Lipuro; Propolipid; Propoven; Recofol; Unifol
  Arms: Propofol

SUMMARY:
The aim of this study is to distinguish possible differences in frequency of delirium after Volatile Induction and Maintenance of Anesthesia and Total Intravenous Anesthesia in case of undeliberate cerebral desaturation during non-cardiac surgery.

DETAILED DESCRIPTION:
The aim of the present study is to investigate whether in non-cardiac surgery the frequency of POD after intraoperative undeliberate cerebral saturation could be modulated by the choice of the anesthetic strategy (Volatile Induction and Maintenance of Anesthesia [VIMA] and Total Intravenous Anesthesia [TIVA]). Based on our previous data we hypothesized that incidence of POD would be lower with VIMA compared to TIVA.

ELIGIBILITY:
Inclusion Criteria:

* class III-IV by physical status classification system of American Society of Anesthesiologist (ASA)
* history of arterial vascular disease (arterial hypertension, myocardial ischemia and/or cerebral vascular disease)
* undergoing elective non-cardiac surgery (hemicolectomy, hernioplasty, laparoscopic cholecystectomy and laparoscopic hysterectomy)

Exclusion Criteria:

* dementia
* stroke or myocardial infarction ≤ 6 months before surgery
* oncological disease of T2-4N3M1 stage

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Regional Cerebral Oxygenation (rSO2) | Continued the entire surgery
Peripheral tissue oxygen saturation (SpO2) | Continued the entire surgery
Non-invasive blood pressure (NIBP) | Continued the entire surgery

SECONDARY OUTCOMES:
Number of Incidences of postoperative delirium (POD) | Baseline, 24h and 48h after surgery
  Applying the Confusion Assessment Method for the ICU (CAM-ICU)
Plasma concentration of S100b protein | Baseline, 24h and 48h after surgery
  S100b protein is the neuronal injury marker

CONTACTS AND LOCATIONS:
Overall Officials: Valery V. Likhvantsev, MD, Prof., Study Chair — Negovsky Reanimatology Research Institute, Moscow, Russia; Oleg A. Grebenchikov, MD, PhD, Study Director — Negovsky Reanimatology Research Institute, Moscow, Russia; Yuri V. Iljin, Principal Investigator — Negovsky Reanimatology Research Institute, Moscow, Russia; Alexander V. Mironenko, MD, PhD, Principal Investigator — Negovsky Reanimatology Research Institute, Moscow, Russia; Yuri V. Skripkin, Principal Investigator — Negovsky Reanimatology Research Institute, Moscow, Russia; Dmitriy B. Selivanov, MD, PhD, Principal Investigator — Hospital Maria Vittoria, Turin, Italy
Locations (1):
- Medical center of the Main Administration for Service to the Diplomatic Corps, Moscow, Russia